CLINICAL TRIAL: NCT03022071
Title: What Works for Whom and How? Mechanisms of Change in Psychotherapy
Brief Title: Mechanisms of Change in Psychotherapy
Acronym: MOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Jan Ivar Røssberg, MD, Professor MD PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: What works for whom and how?
Record Dates: First submitted 2016-11-14; First posted 2017-01-16 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2021-09

CONDITIONS: Depression
Keywords: Cognitive behavior therapy; Psychodynamic therapy; Mediators; Moderators
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy; Psychotherapy, Psychodynamic

STUDY DESIGN:
Intervention Model Description: In this study we want to examine moderators and mediators in two equally effective, well known psychotherapeutic treatments (Psychodynamic and cognitive behavior therapy)
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments will be provided by raters blinded to the randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive behavior therapy (Experimental): The included patients will receive cognitive therapy for depression for 16 weeks and monthly booster sessions up to 28 weeks.
  Interventions: Other: Cognitive behavior therapy
- Psychodynamic psychotherapy (Active Comparator): The included patients will receive time-limited psychodynamic psychotherapy for 28 weeks.
  Interventions: Other: Cognitive behavior therapy

INTERVENTIONS:
Other: Cognitive behavior therapy — In this study we want to compare CBT and PDT and examine whether some patients will benefit from CBT and other from PDT. More specifically we want to examine moderators and mediators for improvement in depressive symptoms in the two interventions arms.
  Other Names: Psychodynamic psychotherapy

SUMMARY:
Background: Major depressive disorder (MDD) is a prevalent psychiatric condition associated with significant disability, mortality and economic burden. MDD is ranked fourth in terms of disease burden as defined by the World Health Organization (2001). Cognitive Behavioral Therapy (CBT) and Psychodynamic Psychotherapy (PDT) are found to be equally effective for patients with depression. However, many patients do not respond sufficiently to treatment and relapse rates are high. To be able to offer individualized treatment, a clinically important question is therefore whether some patients profit more from one of the two therapies. At present little is known on which patient characteristics (moderators) may be associated with differential outcomes of CBT and PDT and through what kind of therapeutic processes and mechanisms (mediators) improvements occur in each therapy mode. There are actually only theoretical assumptions sparsely supported by research findings on what moderates and mediates the treatment effects of CBT and PDT.

Aims: The overall aim of this project is to examine putative moderators and mediators in CBT and PDT and develop more basic knowledge about their impact on outcomes of psychotherapy for patients with MDD.

Methods and study design: The study is a randomized clinical trial. One hundred patients will be randomized to one of two treatment conditions. The patients will be treated over 28 weeks with either CBT (one weekly session over 16 weeks and 3 booster sessions (monthly) during the rest of the 28 week study period) or PDT (one weekly session in 28 weeks). The patients will be evaluated at baseline, during therapy, at the end of therapy, and at follow-up investigations 1 and 3 years after treatment termination. The outcome measures comprise a large range of clinical and process variables, including assessment tools measuring specific preselected putative moderators and mediators.

Discussion: The clinical outcome of this trial may guide clinicians to decide what kind of treatment should be offered the individual patient. Moreover, it will shed light on what kind of mechanisms in psychotherapy that is followed by symptom improvement and increased psychosocial functioning.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18-65 years, with depressive disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV; American Psychiatric Association, 2000) unipolar MDD diagnosis will be included.MINI plus (Sheehan et al., 1998 will be used as assessment tool. Comorbidity is expected to be frequent. Written consent will be obtained from all patients.
* The participants need to have the ability to speak and understand a Scandinavian language, and willingness and ability to give informed consent.

Exclusion Criteria:

* Current or past neurological illness, traumatic brain injury, current alcohol and/or substance dependency disorders, psychotic disorders, developmental disorders, and mental retardation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | Change in scores between baseline and 28 weeks (end of therapy) and change between baseline and one and three year follow-up
  Assessment of depression
Beck Depression Index | Change in scores between baseline and 28 weeks (end of therapy) and change between baseline and one and three year follow-up
  Assessment of depression

SECONDARY OUTCOMES:
Psychodynamic Functioning Scale | Change in scores during therapy and the follow-up periode (one and three years)
  Assesment of dynamic functioning
Beck Cognitive Insight Score | Change in scores during therapy and the follow-up periode (8 weeks, 16 weeks, 28 weeks, 1 year and 3 year follow up)
  Assessment of cognitive insight
Global Assesment of Functioning | Change in scores during therapy and the follow-up periode (one and three years)
  Assessment of global symptoms and functioning
Inventory of Interpersonal Problems | Change in scores during therapy and the follow-up periode (one and three years)
  Measure of interpersonal problems
Reflective functioning - depression | Change in scores during therapy and the follow-up periode (one and three years)
  Assessment of reflective functioning
Dysfunctional Attitude Scale | Change in scores during therapy and the follow-up periode (8 weeks, 16 weeks, 28 weeks, 1 year and 3 year follow up)
  Measure of dysfunctional attitude
Metacognitive questionnaire | Change in scores during therapy and the follow-up periode (8 weeks, 16 weeks, 28 weeks, 1 year and 3 year follow up)
  Assessments of metacognition

OTHER OUTCOMES:
Work and Social Adjustment Scale | Change in scores during therapy and the follow-up periode (8 weeks, 16 weeks, 28 weeks, 1 year and 3 year follow up)
  Assessment of functioning
The Short Form Health Survey | Change in scores during therapy and the follow-up periode (8 weeks, 16 weeks, 28 weeks, 1 year and 3 year follow up)
  Measure of general Health issues
Childhood Trauma Questionnaire | Baseline (inclusion). Moderator of treatment
  Measure of childhood trauma
Severity of Indices of personality Problems | Change in scores during therapy and the follow-up periode (8 weeks, 16 weeks, 28 weeks, 1 year and 3 year follow up)
  Assessments of personality dimensions
Toronto Alexithymia Scale | Change in scores during therapy and the follow-up periode (8 weeks, 16 weeks, 28 weeks, 1 year and 3 year follow up)
  Measures of alexithymia
Rumination respons scale | Change in scores during therapy and the follow-up periode (8 weeks, 16 weeks, 28 weeks, 1 year and 3 year follow up)
  Measures of ruminations
Structural Analysis of Social Behavior | Change in scores during therapy and the follow-up periode (8 weeks, 16 weeks, 28 weeks, 1 year and 3 year follow up)
  Measure social behavior
Experience in Close Relationship Inventory | Change in scores during therapy and the follow-up periode (8 weeks, 16 weeks, 28 weeks, 1 year and 3 year follow up)
  Functioning in Close relations
Patient Health questionnaire | Change in scores during therapy and the follow-up periode (8 weeks, 16 weeks, 28 weeks, 1 year and 3 year follow up)
  Measure anxiety
Hypomani Checlist | Change in scores during therapy and the follow-up periode (one and three years)
  Measures hypomanic symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jan I Røssberg, phD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Malkomsen A, Wilberg T, Bull-Hansen B, Dammen T, Evensen JH, Hummelen B, Lovgren A, Osnes K, Ulberg R, Rossberg JI. Comparative effectiveness of short-term psychodynamic psychotherapy and cognitive behavioral therapy for major depression in psychiatric outpatient clinics: a randomized controlled trial. BMC Psychiatry. 2025 Feb 11;25(1):113. doi: 10.1186/s12888-025-06544-6. PMID 39934737
- [Derived] Malkomsen A, Rossberg JI, Dammen T, Wilberg T, Lovgren A, Ulberg R, Evensen J. How therapists in cognitive behavioral and psychodynamic therapy reflect upon the use of metaphors in therapy: a qualitative study. BMC Psychiatry. 2022 Jun 27;22(1):433. doi: 10.1186/s12888-022-04083-y. PMID 35761306
- [Derived] Malkomsen A, Rossberg JI, Dammen T, Wilberg T, Lovgren A, Ulberg R, Evensen J. Digging down or scratching the surface: how patients use metaphors to describe their experiences of psychotherapy. BMC Psychiatry. 2021 Oct 27;21(1):533. doi: 10.1186/s12888-021-03551-1. PMID 34706691
- [Derived] Rossberg JI, Evensen J, Dammen T, Wilberg T, Klungsoyr O, Jones M, Boen E, Egeland R, Breivik R, Lovgren A, Ulberg R. Mechanisms of change and heterogeneous treatment effects in psychodynamic and cognitive behavioural therapy for patients with depressive disorder: a randomized controlled trial. BMC Psychol. 2021 Jan 22;9(1):11. doi: 10.1186/s40359-021-00517-6. PMID 33482927